CLINICAL TRIAL: NCT04920227
Title: Comparation of CO2 Laser-Assisted Sclerectomy Surgery Combined With Phacoemulsification and CO2 Laser-Assisted Sclerectomy Surgery Alone in the Treatment of Primary Open Angle Glaucoma
Brief Title: Comparation of CLASS Combined With Phacoemulsification and CLASS Alone in the Treatment of Primary Open Angle Glaucoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-528
Record Dates: First submitted 2021-06-01; First posted 2021-06-09 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2020-08

CONDITIONS: Glaucoma, Open-Angle
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Phacoemulsification

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CLASS+PHACO (Experimental): CO2 Laser-Assisted Sclerectomy Surgery combined with phacoemulsification
  Interventions: Procedure: phacoemulsification;
- CLASS (No Intervention): CO2 Laser-Assisted Sclerectomy Surgery

INTERVENTIONS:
Procedure: phacoemulsification; — Group A: class combined with phacoemulsification
  Arms: CLASS+PHACO

SUMMARY:
To compare the effect of intraocular pressure control and the incidence of peripheral anterior synechia between CLASS combined with phacoemulsification and CLASS alone in the treatment of primary open-angle glaucoma

DETAILED DESCRIPTION:
Group A: CO2 Laser-Assisted Sclerectomy Surgery combined with phacoemulsification; Group B: simple CO2 Laser-Assisted Sclerectomy Surgery. The patients were followed up for 1 year. The incidence of peripheral anterior synechia and Intraocular pressure changes at 1 day, 1 week, 1 month, 2 months, 3 months, 6 months and 12 months were observed and compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Primary open-angle glaucoma patients with cataract in our Ophthalmic Center;
* Topical use of hypotensive drugs in the treatment of poor or intolerable intraocular pressure control;
* The patients were aged from 50 to 80 years old, regardless of gender;
* Class operation and phacoemulsification were performed;
* Patients are able and willing to comply with the research guidance and may complete all visits required by the research;
* Informed consent has been signed.

Exclusion Criteria:

* Allergic to any perioperative medication in this study;
* History of ocular trauma;
* Any previous intraocular surgery;
* Angle of the chamber was narrow by angle microscopy (Schaffer grade III and below);
* Patients diagnosed as secondary glaucoma;
* Optic atrophy caused by other reasons;
* The serious complications such as posterior capsule rupture and choroidal hemorrhage occurred during the operation;
* Serious complications of eyes occurred after operation;
* The patient's history indicated that he had severe dysfunction of heart, lung, liver and kidney;
* Women in pregnancy, lactation or planned pregnancy;
* The researchers believe that the patient's condition may put the patient at significant risk, and may confuse the research results.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-09-02 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of peripheral anterior synechia | 1 year
  Incidence of peripheral anterior synechia
Intraocular pressure | 1 year
  Intraocular pressure

CONTACTS AND LOCATIONS:
Overall Officials: Kaijun Wang, MD, Study Director — Eye Center, the 2nd Affiliated Hospital, Medical College of Zhejiang University
Locations (1):
- Eye Center, the 2nd Affiliated Hospital, Medical College of Zhejiang University, Hangzhou, Zhejiang, China